CLINICAL TRIAL: NCT00663442
Title: Dose Response Pharmacogenetic Study of ADHD
Brief Title: Basic and Clinical Research on Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Mark A. Stein Ph.D.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K24-MHO1823
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: ADHD
Keywords: ADHD; side effects; sleep; dopamine; pharmacogenetics
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): OROS methylphenidate 18, 36, 54m placebo in randomized order (except never starting with highest dose)
  Interventions: Drug: OROS methylphenidate

INTERVENTIONS:
Drug: OROS methylphenidate — 18, 36, 54 mg
  Other Names: Concerta

SUMMARY:
Children between 6-17 are evaluated for ADHD and and a blood sample is obtained for DNA extraction. If eligible, they participate in a 4 week, double blind, placebo controlled trial with weekly switches. In randomized order, children receive 18, 36, 54 mg. OROS methylphenidate and placebo. Each week, parent report measures, clinical interviews, and safety assessments are conducted.

Hypothesis: Efficacy and adverse events will be dose dependent. Dopamine Transporter Genotype will predict response

ELIGIBILITY:
Inclusion Criteria:

* 6-17 DSM IV criteria for ADHD Parents willing to complete measures

Exclusion Criteria:

* Mental retardation psychoses seizure disorder

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 1999-12; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
ADHD RS | weekly

SECONDARY OUTCOMES:
CGI-S | weekly
VItal Signs | weekly
Sleep Questionnaire | weekly
Side Effects rating Scale | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Stein, Ph.D., Principal Investigator — Univesity of Illinois at Chicago
Locations (1):
- HALP Clinic, University of Illinois at CHicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Stein MA, Sarampote CS, Waldman ID, Robb AS, Conlon C, Pearl PL, Black DO, Seymour KE, Newcorn JH. A dose-response study of OROS methylphenidate in children with attention-deficit/hyperactivity disorder. Pediatrics. 2003 Nov;112(5):e404. doi: 10.1542/peds.112.5.e404. PMID 14595084
- [Result] Stein MA, Waldman ID, Sarampote CS, Seymour KE, Robb AS, Conlon C, Kim SJ, Cook EH. Dopamine transporter genotype and methylphenidate dose response in children with ADHD. Neuropsychopharmacology. 2005 Jul;30(7):1374-82. doi: 10.1038/sj.npp.1300718. PMID 15827573